CLINICAL TRIAL: NCT02540486
Title: A 12 Week, Parallel, Open-label, Randomized, Multi-center Study Evaluating Use, Safety and Effectiveness of a Web Based Tool vs. Enhanced Usual Therapy of Glargine Titration in T2DM Patients With a 4 Week Safety Extension
Brief Title: Long Acting Insulin Glargine Titration Web Tool (LTHome) vs Enhanced Usual Therapy of Glargine Titration
Acronym: INNOVATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LMC Diabetes & Endocrinology Ltd. (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Principal Investigator, Ronnie Aronson, MD, FRCPC, FACE, LMC Diabetes & Endocrinology Ltd.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INNOVATE
Record Dates: First submitted 2015-08-21; First posted 2015-09-04 (Estimated); Last update posted 2015-09-04 (Estimated); Status verified 2015-09

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 diabetes; T2DM
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LTHome web tool (Experimental): The long-acting insulin glargine titration web tool (LTHome) will provide insulin glargine titration suggestions based on user inputted blood glucose readings.
  Interventions: Other: Long-acting insulin glargine titration web tool (LTHome); Other: Diabetes Education
- Enhanced Usual Therapy (EUT) (Active Comparator): The Enhanced Usual Therapy arm will receive insulin glargine titration instructions that are the usual therapy provided by the physician/HCP, in addition to diabetes education.
  Interventions: Other: Diabetes Education

INTERVENTIONS:
Other: Long-acting insulin glargine titration web tool (LTHome) — The LTHome study arm will receive insulin glargine titration instructions from the LTHome web-based tool
  Arms: LTHome web tool
Other: Diabetes Education — Individual diabetes education, detailed instructions on the use of the blood glucose monitor and unlimited availability of blood glucose monitoring supplies.

SUMMARY:
Evaluating patients with type 2 diabetes either starting once daily basal insulin or requiring increased basal titrations in order to compare the LTHome web based tool with the usual standard of practice for insulin glargine dosing adjustment.

DETAILED DESCRIPTION:
INNOVATE is a 12 week, parallel, open-label, randomized, multi-center study evaluating use, safety and effectiveness of a web based tool (LTHome) vs. enhanced usual therapy (EUT) of glargine titration in T2DM patients.

The primary objective of this study is to compare the effectiveness LTHome versus EUT of glargine titration in people with T2DM patients on basal insulin not meeting local targets or patients requiring basal initiation. Success will be measured by the percentage of subjects reaching Canadian Diabetes Association (CDA) guideline targets.

The efficacy objective is to demonstrate that the percentage (%) of subjects to reach FPG target by titration of insulin glargine using the LTHome tool with dose adjustment advice is not inferior to the % of subjects to reach FPG target using Enhanced Usual Therapy glargine titration during study participation (LTHome vs. EUT treatments).

The secondary objectives of this study are to assess safety, effectiveness, satisfaction and adherence of LTHome use versus Enhanced Usual Therapy glargine titration.

ELIGIBILITY:
Inclusion Criteria:

* Patient with type 2 diabetes mellitus (T2DM) between 18 and 75 years old (inclusively) with BMI ≤ 45 kg/m2.
* Signed written informed consent
* Patients scheduled to: initiate basal insulin treatment or increase their dose of current basal insulin therapy, independently of study participation, because of :

  • inadequate blood glucose control
* If on basal therapy at screening, must be using a stable dose of insulin glargine x 1 week prior to randomization
* Patients with poor blood glucose control defined by:

  * HbA1c level between > 7% at screening AND
  * mean FPG > 7 mmol/l as determined by most recent self-measured blood glucose in 3 of 7 days prior to randomization
* Patients proficient in computer literacy
* Patient is able and willing to monitor glucose with a home glucose monitor, and consistently record his/her blood glucose and insulin doses in a patient diary/web tool.

Exclusion Criteria:

* Any technical/administrative reason that makes it impossible to include the patient in the study, including closing enrollment due to full enrollment
* Patient who has previously participated in any clinical trial investigating the LTHome algorithm
* Patient who withdraws consent during screening (starting from signed informed consent form)
* Use of systemic steroids in the last 90 days
* Conditions/situations:

  * Patients with short life expectancy (less than 1 year)
  * Type 1 diabetes mellitus
  * Patients with conditions/concomitant diseases making them non-evaluable for the primary efficacy endpoint
  * Clinically significant cardiac disease, retinopathy, hepatic, renal dysfunction or relevant other major diseases as determined by Principal Investigator or designee.
  * Unstable oral antihyperglycemic drugs and/or Glucagon-Like Peptide Receptor (GLP-1R) Agonists therapy during the 4 week period prior to screening
  * Impossibility to meet specific protocol requirements (e.g. ability to perform blood glucose measurements, manage their own insulin glargine administration or deemed unlikely to safely manage insulin dosage on guidance by their HCP)
  * Patient is a primary relative of the Investigator or any Sub-Investigator, research assistant, pharmacist, study coordinator, or other staff or is directly involved in the conduct of the protocol
  * Patients with hypoglycemia unawareness, severe hypoglycemic episode in the last 90 days or hospitalization (for any reason) in the last 30 days
  * Cognitive disorder, dementia or any neurologic disorder, that would affect patient's ability to participate in the study, or patients who have no legal capacity or are under guardianship
* Pregnant or breastfeeding women, or women of child-bearing potential not protected by highly effective method(s) of birth control (as defined in the informed consent form and/or in a local protocol addendum) and who are unwilling or unable to be tested for pregnancy.
* Patients who are using, or need to start using, mealtime (Bolus) insulin during the timeframe of the study.
* Night shift workers

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2013-12; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects reaching fasting plasma glucose (FPG) target | 12 weeks
  The primary outcome is defined as all of the following
  * At least 4 out of 7 FPG readings done within a 10 day period are within the target range of 5-7.2 mmol/L
  * Mean glucose for three consecutive prior FPG values is between 5-7.2 mmol/L
  * There is no severe hypoglycemia during the 7-10 day period (Severe hypoglycemia is defined as third party intervention in management of the hypoglycemia).

SECONDARY OUTCOMES:
Number of days to first reach fasting plasma glucose target | 12 weeks
  The number of days in the study until the first day the target is reached.
Number of days in target range after reaching fasting plasma glucose target | 12 weeks
  The number of days after reaching target where the FPG was between 5.0 and 7.2 mmol/L (inclusive)
Fasting plasma glucose | 12 weeks
  Fasting plasma glucose values over the entire study period will be summarized by mean and standard deviation
Hemoglobin A1c (HbA1c) | 12 weeks
  The change in HbA1c will be evaluated as an expression of overall glycemic control in the two treatment arms and compared.
Rate of documented hypoglycemia in subjects that reach target | 12 weeks
Rate of documented hypoglycemia in subjects that do not reach target | 12 weeks
Proportion of all patients with hypoglycemia | 12 weeks
  A summary of any hypoglycemia, severe hypoglycemia, nocturnal hypoglycemia, day-time hypoglycemia, symptomatic hypoglycemia, probable symptomatic hypoglycemia, and asymptomatic hypoglycemia will be summarized
Frequency of contact with physician/HCP | 12 weeks
  The number of times subjects contacted their physician/HCP during the study
Diabetes Treatment Satisfaction Questionnaire (DTSQ) | 12 weeks
  A questionnaire to assess subject's overall satisfaction with their diabetes treatment
Hypoglycemia Fear Survey (HFS) | 12 weeks
  A questionnaire to assess the subject's behaviours to avoid hypoglycemia and to measure the subjects' worries about hypoglycemia and its consequences
WHO-5 Well-Being Index | 12 weeks
  A questionnaire to measure emotional well-being to screening for likely depression in subjects with diabetes
Diabetes Distress Scale | 12 weeks
  A questionnaire to assess diabetes-related emotional distress
LTHome Patient Satisfaction Survey | 12 weeks
  LTHome arm only; a questionnaire to measure satisfaction of the use of the LTHome
Number of days subjects self-monitored their fasting plasma glucose | 12 weeks
Number of dose recommendations prior to reaching target - LTHome only | 12 weeks
Number of dose recommendations after target is reached - LTHome only | 12 weeks
Number of days insulin glargine was taken - LTHome only | 12 weeks
Reasons for disregarding LTHome advice - LTHome only | 12 weeks
  A summary of the reasons that subjects gave for not taking the insulin glargine dose recommendation given by the LTHome web tool when the recommendation was not followed
Adverse events | 12 weeks
Serious adverse events | 12 weeks

OTHER OUTCOMES:
Body weight (kg) | 12 weeks
List of concomitant medications initiated after randomization | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ronnie Aronson, MD, Principal Investigator — LMC Diabetes & Endocrinology Ltd.
Locations (1):
- LMC Diabetes & Endocrinology, Toronto, Ontario, Canada

REFERENCES:
- [Background] Workgroup on Hypoglycemia, American Diabetes Association. Defining and reporting hypoglycemia in diabetes: a report from the American Diabetes Association Workgroup on Hypoglycemia. Diabetes Care. 2005 May;28(5):1245-9. doi: 10.2337/diacare.28.5.1245. No abstract available. PMID 15855602
- [Background] Strange P. Treat-to-target insulin titration algorithms when initiating long or intermediate acting insulin in type 2 diabetes. J Diabetes Sci Technol. 2007 Jul;1(4):540-8. doi: 10.1177/193229680700100412. PMID 19885117
- [Background] Morrison F, Shubina M, Turchin A. Encounter frequency and serum glucose level, blood pressure, and cholesterol level control in patients with diabetes mellitus. Arch Intern Med. 2011 Sep 26;171(17):1542-50. doi: 10.1001/archinternmed.2011.400. PMID 21949161
- [Background] Nathan DM, Buse JB, Davidson MB, Ferrannini E, Holman RR, Sherwin R, Zinman B; American Diabetes Association; European Association for Study of Diabetes. Medical management of hyperglycemia in type 2 diabetes: a consensus algorithm for the initiation and adjustment of therapy: a consensus statement of the American Diabetes Association and the European Association for the Study of Diabetes. Diabetes Care. 2009 Jan;32(1):193-203. doi: 10.2337/dc08-9025. Epub 2008 Oct 22. PMID 18945920
- [Background] Cryer PE. Hypoglycaemia: the limiting factor in the glycaemic management of Type I and Type II diabetes. Diabetologia. 2002 Jul;45(7):937-48. doi: 10.1007/s00125-002-0822-9. Epub 2002 Apr 26. PMID 12136392
- [Background] Zammitt NN, Frier BM. Hypoglycemia in type 2 diabetes: pathophysiology, frequency, and effects of different treatment modalities. Diabetes Care. 2005 Dec;28(12):2948-61. doi: 10.2337/diacare.28.12.2948. No abstract available. PMID 16306561
- [Background] Briscoe VJ, Davis SN. Hypoglycemia in type 1 and type 2 diabetes: physiology, pathophysiology, and management. Clinical Diabetes 24(3): 115-121, 2006.
- [Background] Seaquist ER, Miller ME, Bonds DE, Feinglos M, Goff DC Jr, Peterson K, Senior P; ACCORD Investigators. The impact of frequent and unrecognized hypoglycemia on mortality in the ACCORD study. Diabetes Care. 2012 Feb;35(2):409-14. doi: 10.2337/dc11-0996. Epub 2011 Dec 16. PMID 22179956
- [Background] Swinnen SG, Hoekstra JB, DeVries JH. Insulin therapy for type 2 diabetes. Diabetes Care. 2009 Nov;32 Suppl 2(Suppl 2):S253-9. doi: 10.2337/dc09-S318. No abstract available. PMID 19875560
- [Background] Boussageon R, Bejan-Angoulvant T, Saadatian-Elahi M, Lafont S, Bergeonneau C, Kassai B, Erpeldinger S, Wright JM, Gueyffier F, Cornu C. Effect of intensive glucose lowering treatment on all cause mortality, cardiovascular death, and microvascular events in type 2 diabetes: meta-analysis of randomised controlled trials. BMJ. 2011 Jul 26;343:d4169. doi: 10.1136/bmj.d4169. PMID 21791495
- [Background] Epidemiology of severe hypoglycemia in the diabetes control and complications trial. The DCCT Research Group. Am J Med. 1991 Apr;90(4):450-9. PMID 2012085
- [Background] Bradley C, Plowright R, Stewart J, Valentine J, Witthaus E. The Diabetes Treatment Satisfaction Questionnaire change version (DTSQc) evaluated in insulin glargine trials shows greater responsiveness to improvements than the original DTSQ. Health Qual Life Outcomes. 2007 Oct 10;5:57. doi: 10.1186/1477-7525-5-57. PMID 17927832
- [Background] Cox DJ, Irvine A, Gonder-Frederick L, Nowacek G, Butterfield J. Fear of hypoglycemia: quantification, validation, and utilization. Diabetes Care. 1987 Sep-Oct;10(5):617-21. doi: 10.2337/diacare.10.5.617. PMID 3677982
- [Background] Hajos TR, Pouwer F, Skovlund SE, Den Oudsten BL, Geelhoed-Duijvestijn PH, Tack CJ, Snoek FJ. Psychometric and screening properties of the WHO-5 well-being index in adult outpatients with Type 1 or Type 2 diabetes mellitus. Diabet Med. 2013 Feb;30(2):e63-9. doi: 10.1111/dme.12040. PMID 23072401
- [Background] Polonsky WH, Fisher L, Earles J, Dudl RJ, Lees J, Mullan J, Jackson RA. Assessing psychosocial distress in diabetes: development of the diabetes distress scale. Diabetes Care. 2005 Mar;28(3):626-31. doi: 10.2337/diacare.28.3.626. PMID 15735199
- [Background] Petznick A. Insulin management of type 2 diabetes mellitus. Am Fam Physician. 2011 Jul 15;84(2):183-90. PMID 21766768
- [Background] Canadian Diabetes Association Clinical Practice Guidelines Expert Committee; Cheng AY. Canadian Diabetes Association 2013 clinical practice guidelines for the prevention and management of diabetes in Canada. Introduction. Can J Diabetes. 2013 Apr;37 Suppl 1:S1-3. doi: 10.1016/j.jcjd.2013.01.009. Epub 2013 Mar 26. No abstract available. PMID 24070926